CLINICAL TRIAL: NCT04409587
Title: Basal Insulin Glycemic ControL With DEglugec vs Aspart Via Pump: A Comparison of Insulin Degludec to Continuous Subcutaneous Infusion of Insulin Aspart for Basal Insulin Delivery in Type 1 Diabetes
Brief Title: Basal Insulin Glycemic ControL With DEglugec vs Aspart Via Pump
Acronym: BIG LEAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mountain Diabetes and Endocrine Center (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MDEC2018
Record Dates: First submitted 2018-07-30; First posted 2020-06-01 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Continuous Glucose Monitoring; CGM; Continuous Subcutaneous Insulin Infusion
MeSH Terms: interventions — Insulin Aspart; insulin degludec

STUDY DESIGN:
Intervention Model Description: This will be a randomized, cross-over, open label, single-center study consisting of a 20 week period on each of two basal insulin delivery methods, both in combination with insulin aspart with boluses taken by insulin pump. Each 20 week period will consist of a 4 week insulin optimization period for titration of basal and bolus insulin doses, followed by a 16 week maintenance period. The final 2 weeks of the maintenance period during each treatment arm will be used for endpoint data collection. The treatment sequence will occur in random order. The study population will include patients with type 1 diabetes with good baseline glycemic control who are experienced in the use of both Continuous Subcutaneous Insulin Infusion and Continuous Glucose Monitor; the cross-over design allows each subject to serve as his or her own control.
Masking Description: This is an unblinded study as the two basal insulin delivery methods (degludec via injection vs. aspart via CSII) cannot be blinded. One group of patients will first use degludec for 20 weeks then switch to CSII for 20 weeks. As all eligible patients who sign the IRB consent form are identified, a random number will be generated to determine the treatment with which they begin first. The other group of patients will start with CSII and after 20 weeks switch to Tresiba for 20 weeks. Randomization sequence will be determined by computerized randomization program. All patients will receive both treatments unless they drop out. Dropouts are unlikely since the participants are all regular continuing patients of the site's clinical practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NovoLog®-only (No Intervention): In the aspart-Only group, the subject will only take aspart through the their pump. This study population will have an established expertise in diabetes self-management with previous knowledge of insulin pump therapy and Dexcom Continuous Glucose Monitoring (CGM). Allowing the subjects to use their insulin pumps for bolus insulin delivery, as they are accustomed, will minimize the chances of skipping meal boluses and correction doses. Aspart is put into their pump and delivered to their body through a small tube placed under your skin. In this NovoLog®-only treatment group, the subject will take aspart with each meal while your pump also gives you a slow, continuous dose of aspart for basal insulin. This treatment group is very similar (or even identical) to the treatment the subject was receiving prior to starting the study.
- Novolog® and Tresiba® Group (Active Comparator): This study population will have an expertise in diabetes self-management with their insulin pump and Dexcom CGM. In the Novolog® and Tresiba® group, the subject will still take aspart via their pump for meals and correction boluses, but they will reduce the slow trickle (basal insulin) programmed in their pump to almost zero. Instead of receiving their normal basal insulin via CSII, the subject will injected degludec once or twice daily from an insulin pen for your basal insulin.
  Interventions: Drug: Aspart

INTERVENTIONS:
Drug: Aspart — A population of well controlled patients with type 1 diabetes who are experienced in the use of both Continuous Subcutaneous Insulin Infusion (CSII) and Continuous Glucose Monitor (CGM) was chosen in order to assess the effect of the change in glycemic profile using two different methods of basal insulin delivery. Allowing the subjects to use their insulin pumps for bolus insulin delivery, as they are accustomed, will minimize the chances of skipping meal boluses and correction doses.
  Replacing basal insulin delivery by CSII with a single daily injection of degludec will add minimal, if any, treatment burden which will be offset by potential therapeutic benefits. These benefits include the potential for reduced glycemic variability and the elimination of the risk of hyperglycemia and DKA with basal insulin interruption which can occur with infusion set occlusion or disgorging inherent to Continuous Subcutaneous Insulin Infusion.
  Other Names: Degludec
  Arms: Novolog® and Tresiba® Group

SUMMARY:
The purpose of this investigator-initiated trial is to compare the effect of a daily injection of insulin degludec vs. basal insulin delivery via Continuous Subcutaneous Insulin Infusion (CSII), both in combination with bolus insulin delivery via the patient's usual insulin pump with insulin aspart, on glycemic variability, overall blood glucose control and incidence of hypoglycemia, all assessed by continuous glucose monitor (CGM), as well as patient satisfaction, in patients with type 1 diabetes currently using CSII.

DETAILED DESCRIPTION:
The primary objective of this trial is to determine whether insulin degludec will provide an equally stable and consistent basal glycemic profile with lower glycemic variability as determined by Continuous Glucose Monitoring compared to insulin aspart delivered by Continuous Subcutaneous Insulin Infusion in patients with type 1 diabetes experienced in use of insulin pump therapy. Specifically, this study will determine if the percent time in the target glycemic range (70 to 180 mg/dl) by Continuous Glucose Monitoring is superior using insulin degludec than continuously infused insulin aspart, and if degludec is associated with lower glucose variability as assessed by the standard deviation (SD) of the mean daily glucose by Continuous Glucose Monitoring. Particular attention will be given to the nocturnal glucose profile (from midnight to 6 am) which most closely reflects basal insulin action as it is typically the time of day least affected by bolus insulin, food intake or exercise. Quality of life questionnaires regarding treatment preference will be used to capture patient preference for method of basal insulin delivery.

RESEARCH DESIGN AND METHODS

Study hypothesis:

It is anticipated, based on the low glycemic variability of insulin degludec shown in glucose clamp studies and seen in clinical practice, that insulin degludec will provide more stable 24 hour basal insulin action than insulin aspart by Continuous Subcutaneous Insulin Infusion (CSII) in patients with type 1 diabetes.

Primary endpoint:

Percent time in euglycemia (BG 70 to 180 mg/dl) by Continuous Glucose Monitoring (CGM) during the final 14 days of each treatment period during steady state (with basal insulin delivery as either one daily injection of insulin degludec or as insulin aspart via CSII).

Study type:

This will be a randomized, cross-over, open label, single-center study consisting of a 20 week period on each of two basal insulin delivery methods, both in combination with insulin aspart with boluses taken by insulin pump. Each 20 week period will consist of a 4 week insulin optimization period for titration of basal and bolus insulin doses, followed by a 16 week maintenance period. The final 2 weeks of the maintenance period during each treatment arm will be used for endpoint data collection. The treatment sequence will occur in random order. The study population will include patients with type 1 diabetes with good baseline glycemic control who are experienced in the use of both CSII and CGM; the cross-over design allows each subject to serve as his or her own control.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients > 18 years of age with type 1 diabetes using CSII with any pump for > 12 months.
2. Females must be using adequate contraception, defined as oral contraceptive pill, barrier method of contraception, or surgical method (tubal ligation or hysterectomy).
3. Good glycemic control (HbA1c < 8.0%).
4. Patients are experienced in carbohydrate counting, evidenced by pump downloads showing frequent meal boluses with realistic carbohydrate entries, few over-rides of the pump bolus calculator, few to no omitted boluses (at least 3 boluses per day), and post-meal glucose levels generally below 200 mg/dl indicating accurate carbohydrate assessment.
5. Patients are regular (>85% of time) users of the Dexcom G5 or G6 CGM.
6. Pump download confirms correct use of insulin pump features, including appropriate use of bolus calculator with minimal overrides, entering carbohydrate content of meals, at least 3 boluses taken per day, appropriate use of correction boluses, and infusion set changes every 2 to 3 days.
7. No serious comorbidities including: retinopathy requiring active intervention, eGFR < 30, CV event within the previous 6 months, active malignancy with ongoing treatment, any condition requiring chronic use of systemic glucocorticoids, or any other condition which in the opinion of the investigator would interfere with the subject's ability to comply with the study protocol or acutely affect insulin requirements.
8. Able to comply with study protocol.
9. Ability to provide written informed consent prior to any study-related procedures.

   -

Exclusion Criteria:

1. Subjects with type 2 diabetes.
2. Subjects with HbA1c > 8.0%
3. Subjects not using CSII and CGM (ie, on MDI)
4. Subjects inexperienced in the use of CSII, or whose pump download shows poor utilization of bolus calculator features, ie fewer than 2 boluses per day, lack of correction boluses, frequent overrides of the recommended boluses, unrealistic carbohydrate entries (suggestive of under-bolusing), not changing infusion set at least every 3 days, or other evidence of poor insulin pump usage.
5. Subjects inexperienced in or not regular users (>85% of time) of Dexcom G5 or G6 CGM
6. Subjects who are using a Medtronic pump with low blood glucose suspend who are unwilling to use the Dexcom CGM or to disengage the low blood glucose suspend feature of the pump.
7. Use of any other CGM than Dexcom G5 or G6.
8. Serious concomitant illness.
9. Females unwilling to use adequate contraception, intending to become pregnant, or breastfeeding.
10. Known or suspected allergy to study products, their excipients or related products.
11. Previous participation in this trial. Note: subjects who screen fail because of A1c may rescreen once if, in the opinion of the investigator, the HbA1c was explainable (ie, recent steroid injection or illness, etc) and atypical for the subject.
12. Hypoglycemic unawareness.
13. Episode of severe hypoglycemia (requiring assistance for treatment) within the previous 90 days.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Percent time in euglycemia (BG 70 to 180 mg/dl) by CGM | 46 weeks
  Percent time in euglycemia (BG 70 to 180 mg/dl) by CGM during the final 14 days of each treatment period during steady state (with basal insulin delivery as either one daily injection of insulin degludec or as insulin aspart via CSII)

SECONDARY OUTCOMES:
Standard Deviation (SD) of blood glucose by CGM for two week period | 46 weeks
  SD of interstitial fluid glucose by CGM for 2 week period during each basal insulin delivery method. (Note: because the Dexcom Platinum G5 CGM is currently only FDA approved for 7 days of use, two contiguous CGM periods using 2 sensors, each for 7 days, will be performed to capture 2 weeks of continuous CGM data.) Dexcom G6 is approved by FDA for 10 days of use so 2 sensors will be used during the CGM periods.
SD of blood glucose by CGM during the nocturnal period | 46 weeks
  SD of blood glucose by CGM during the nocturnal period (midnight to 6 am) during each basal insulin delivery method
Percent time in hypoglycemia by CGM | 46 weeks
  Percent time in hypoglycemia by CGM, captured at 2 levels of hypoglycemia: BG < 54 mg/dl (level 2) and BG 55-69 mg/dl (level 1), for each basal insulin treatment.
Percent time in normoglycemia | 46 weeks
  Percent time in normoglycemia (BG 70 to 140 mg/dl) by CGM during each basal treatment period.
Time to recovery from level 2 hypoglycemia | 46 weeks
  Time to recovery from level 2 hypoglycemia (BG >70 with resolution of symptoms) on each treatment. If a second event (BG < 70 mg/dl) occurs within 60 minutes of a previous hypoglycemic event, this will be considered part of the same hypoglycemic episode.
Patient satisfaction | 46 weeks
  Patient satisfaction by TRIM-D questionnaires with each basal insulin treatment.
Patient satisfaction | 46 weeks
  Patient satisfaction by TRIM-DD questionnaires with each basal insulin treatment.
HbA1c | 46 weeks
  HbA1c after 20 weeks of each basal insulin treatment.
Total daily insulin dosage | 46 weeks
  Total daily insulin dose, total basal insulin dose, and total bolus insulin dose on each treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Mountain Diabetes and Endocrine Center, Asheville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and statistical analysis will be available to any researcher with appropriate request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: post study, up to 5 years
Access Criteria: email principal investigator

REFERENCES:
- [Result] Misso ML, Egberts KJ, Page M, O'Connor D, Shaw J. Continuous subcutaneous insulin infusion (CSII) versus multiple insulin injections for type 1 diabetes mellitus. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD005103. doi: 10.1002/14651858.CD005103.pub2. PMID 20091571
- [Result] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Result] Heise T, Hermanski L, Nosek L, Feldman A, Rasmussen S, Haahr H. Insulin degludec: four times lower pharmacodynamic variability than insulin glargine under steady-state conditions in type 1 diabetes. Diabetes Obes Metab. 2012 Sep;14(9):859-64. doi: 10.1111/j.1463-1326.2012.01627.x. Epub 2012 Jun 7. PMID 22594461
- [Result] Lane W, Bailey TS, Gerety G, Gumprecht J, Philis-Tsimikas A, Hansen CT, Nielsen TSS, Warren M; Group Information; SWITCH 1. Effect of Insulin Degludec vs Insulin Glargine U100 on Hypoglycemia in Patients With Type 1 Diabetes: The SWITCH 1 Randomized Clinical Trial. JAMA. 2017 Jul 4;318(1):33-44. doi: 10.1001/jama.2017.7115. PMID 28672316
- [Result] Bergenstal RM, Garg S, Weinzimer SA, Buckingham BA, Bode BW, Tamborlane WV, Kaufman FR. Safety of a Hybrid Closed-Loop Insulin Delivery System in Patients With Type 1 Diabetes. JAMA. 2016 Oct 4;316(13):1407-1408. doi: 10.1001/jama.2016.11708. No abstract available. PMID 27629148
- [Result] Novo Nordisk. (2015). TRESIBA® (insulin degludec injection) Label. 28-29
- [Result] Novo Nordisk. (2000). NovoLog (insulin aspart [rDNA origin]) injection label. 21-22
- See also: Hauzenber JR et al. Diab Technol Therapeutics 2017 — http://online.liebertpub.com/doi/full/10.1089/DIA.2017.0175

DOCUMENTS (1):
  • Study Protocol (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT04409587/Prot_000.pdf